CLINICAL TRIAL: NCT06934655
Title: Early Re-Initiation of Semaglutide Post Sleeve Gastrectomy in Youth
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Alaina P. Vidmar, MD, Associate Professor of Pediatrics, Director of Obesity Medicine and Bariatric Surgery, Children's Hospital Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHLA-18-00416
Record Dates: First submitted 2025-03-24; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Pediatric Obesity; Metabolic and Bariatric Surgery; Semaglutide
MeSH Terms: conditions — Pediatric Obesity | interventions — semaglutide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Care (No Intervention): Standard of care following bariatric surgery. No Reinitiation of obesity optimizing medications.
- Early reinitiation (Experimental): Early Reinitiation of semaglutide at 2 weeks after bariatric surgery per standard titration starting at 0.25 mg weekly and titrating to 2.4 mg weekly
  Interventions: Drug: Semaglutide 2.4 mg

INTERVENTIONS:
Drug: Semaglutide 2.4 mg — The dosing regimen will follow standard titration protocols, starting with a dose of 0.25 mg weekly for the first month, with gradual increases in dosage each month to a target dose of 2.4 mg weekly by the fifth month. To minimize the potential for side effects impacting daily activities, youth in the semaglutide group will be instructed to administer the medication weekly on Fridays.
  Other Names: Wegovy
  Arms: Early reinitiation

SUMMARY:
This is a Phase 3a, randomized, parallel-controlled trial designed to compare the early re-initiation of semaglutide, starting two weeks after sleeve gastrectomy, to standard care (no pharmacotherapy following surgery). The trial will involve 150 youth with severe obesity who have been on semaglutide 2.4 mg weekly for at least 3 months prior to surgery. Participants will be randomized to either (1) semaglutide 2.4 mg weekly or (2) standard care for 24 months. Primary, secondary, and tertiary outcomes will be assessed at multiple time points: 1-month, day of surgery, and 1-, 3-, 6-, 9-, 12-, 18-, and 24-months postoperatively. We hypothesize that early re-initiation of semaglutide will be safe, well-tolerated, and lead to greater improvements in obesity, cardiometabolic risk, and eating behaviors.

DETAILED DESCRIPTION:
Study Design: Phase 3a Randomized Controlled Trial of Early Re-initiation of Semaglutide After Sleeve Gastrectomy in Youth with Severe Obesity

Study Type: Interventional (Clinical Trial)

Study Phase: Phase 3a

Allocation: Randomized

Intervention Model: Parallel Assignment

Primary Purpose: Treatment

Participants: Estimated Enrollment - 150 participants

Population:

Youth aged [12-18] with severe obesity who have:

Undergone sleeve gastrectomy

Been on semaglutide 2.4 mg weekly for at least 3 months prior to surgery

Intervention Arms:

Arm 1: Semaglutide Re-initiation Group

Semaglutide 2.4 mg once weekly

Re-initiated 2 weeks after sleeve gastrectomy

Continued for 24 months postoperatively

Arm 2: Standard Care Group

No pharmacotherapy postoperatively

Routine postoperative clinical follow-up for 24 months

Assessment Time Points:

Preoperative Assessments:

1 month before surgery

Day of surgery

Postoperative Assessments:

1 month

3 months

6 months

9 months

12 months

18 months

24 months

Outcomes:

Primary Outcome:

Change in BMI or BMI z-score from baseline to 24 months

Secondary Outcomes:

Safety and tolerability of early semaglutide re-initiation

Changes in weight and waist circumference

Changes in cardiometabolic markers (e.g., HbA1c, lipids, blood pressure)

Tertiary Outcomes:

Changes in eating behaviors

Quality of life assessments

Adherence and persistence with medication

Rate of postoperative complications

ELIGIBILITY:
Inclusion Criteria:

* ages 12 to 18 years
* Tanner stage 3 or higher
* severe obesity (defined as a BMI greater than 35 kg/m2 or BMI ≥140% of the 95th percentile)
* currently undergoing primary surgical weight loss through the pediatric bariatric surgery pathway at Children's Hospital Los Angeles
* be willing to have blood collected before and after surgical procedure at defined points
* be willing to have clinical data entered into a prospective database; 8) presence of a consenting caregiver
* be taking semaglutide 2.4 mg weekly as part of their routine medical care prior to surgery as part of their obesity treatment program, apart from any planned surgical procedure.

Exclusion Criteria:

* have a previous diagnosis of type 1 diabetes
* taking any medications known to influence body composition or prevent weight loss or promote weight gain (e.g. prednisone)
* have been diagnosed with syndromes or diseases that may influence the postoperative course (e.g., Cushing syndrome, Down syndrome, Prader Willi Syndrome)
* have significant comorbid medical conditions necessitating frequent hospitalization that may require interruption of medications and/or that would make early re-initiation of semaglutide unsafe due to the other medical comorbidities
* refuse to comply with eligibility criteria.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2030-11-01 (Estimated); Study Completion 2033-11-01 (Estimated)

PRIMARY OUTCOMES:
Percent Body Mass Index | From enrollment to the end of the end of the study at 24 months
  Percent Body Mass Index (%BMI) is calculated as the participant's BMI at each assessment time point expressed as a percentage of the 95th percentile BMI for age and sex, based on CDC growth charts. This metric is commonly used in pediatric populations to more accurately reflect degrees of obesity in youth, particularly at the upper end of the BMI distribution where standard BMI z-scores may lose sensitivity.
  Calculation Formula:
  %BMI = (Participant's BMI / 95th percentile BMI for age and sex) × 100
  Type (continuous)
  Units (Percent)
  Justification:
  %BMI is used as a more precise and interpretable measure of adiposity in children and adolescents with severe obesity. It allows for consistent tracking of obesity severity and treatment response over time, even in populations whose BMI values significantly exceed the 95th percentile.

SECONDARY OUTCOMES:
Modified percent time in range | From enrollment to the end of the study period at 24 months
  Modified Percent Time in Range (TIR) is defined as the proportion of time a participant's blood glucose levels fall within the target glycemic range of 70-140 mg/dL, as measured by continuous glucose monitoring (CGM). This narrower range is selected to reflect more stringent glycemic control goals for youth with type 2 diabetes and to better capture early intervention effects on glucose regulation. TIR is expressed as a percentage of total monitored time.
  Calculation:
  TIR (%) = (Time within 70-140 mg/dL / Total monitored time) × 100 Data on time above range (TAR; >140 mg/dL) and time below range (TBR; <70 mg/dL) may also be collected as exploratory or secondary metrics.
  Type:
  Continuous
  Units:
  Percent (%)

OTHER OUTCOMES:
Eating in the absence of hunger | Month 24 compared to baseline
  This outcome measures Eating in the Absence of Hunger (EAH) using a validated laboratory-based protocol designed to assess non-homeostatic eating behaviors in children and adolescents. EAH is defined as the intake of palatable foods when an individual is physically satiated, capturing susceptibility to external food cues and emotional or hedonic eating. During the lab experiment, participants are first provided with a standardized meal designed to achieve satiety. Following a brief rest period, participants are then given free access to a variety of palatable snack foods (e.g., chips, cookies, candy) in a controlled setting, with no time pressure and no encouragement to eat. The total caloric intake during this period is measured and recorded.
  Type:
  Continuous
  Units:
  Kilocalories (kcal) consumed during the EAH protocol

CONTACTS AND LOCATIONS:
Overall Officials: Alaina Vidmar, MD, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant Data that underlie the results reported in this study will be shared after de-identification. This includes all data collected at the individual level for primary, secondary, and exploratory outcomes.
  Types of IPD to be Shared:
  De-identified demographic and baseline characteristics
  Primary outcome data
  Secondary outcome data
  Adherence and safety data
  How to Request Access:
  Researchers should contact the principal investigator through the University of Southern California institutional repository. Specific details on data availability and request procedures will be posted with the publication of study findings.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD will be made available no later than 24 months after study completion (defined as final follow-up visit for the last participant) and will remain available for up to 5 years following publication of the primary results.
Access Criteria: Data will be shared with qualified researchers upon request for the purpose of academic research. Requests must include a methodologically sound proposal and will be reviewed by the study's data access committee. All requestors must agree to a data use agreement to ensure participant confidentiality and appropriate data handling.